CLINICAL TRIAL: NCT01178073
Title: AMBITION: A Randomised, Multicenter Study of First-Line Ambrisentan and Tadalafil Combination Therapy in Subjects With Pulmonary Arterial Hypertension (PAH)
Brief Title: A Study of First-Line Ambrisentan and Tadalafil Combination Therapy in Subjects With Pulmonary Arterial Hypertension (PAH)
Acronym: AMBITION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112565
Record Dates: First submitted 2010-07-15; First posted 2010-08-09 (Estimated); Results first posted 2015-04-28 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary Arterial Hypertension; Ambrisentan; Sponsor Rest of World: GSK; Tadalafil; PAH; Sponsor US: Gilead
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — ambrisentan; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Combination ambrisentan + tadalafil (Active Comparator): ambrisentan + tadalafil
  Interventions: Drug: ambrisentan; Drug: tadalafil
- Monotherapy ambrisentan (Active Comparator): ambrisentan
  Interventions: Drug: ambrisentan
- Monotherapy tadalafil (Active Comparator): tadalafil
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: ambrisentan — ambrisentan (target dose: 10mg)
  Arms: Combination ambrisentan + tadalafil; Monotherapy ambrisentan
Drug: tadalafil — tadalafil (target dose: 40mg)
  Arms: Combination ambrisentan + tadalafil; Monotherapy tadalafil

SUMMARY:
The purpose of this study is to compare the two treatment strategies; first-line combination therapy (ambrisentan and tadalafil) versus first-line monotherapy (ambrisentan or tadalafil) in subjects with Pulmonary Arterial Hypertension. This will be assessed by time to the first clinical failure event.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of Pulmonary Arterial Hypertension (PAH) due to the following:

  a. idiopathic or heritable PAH b. PAH associated with: i. connective tissue disease (e.g., limited scleroderma, diffuse scleroderma, mixed connective tissue disease, systemic lupus erythematosus, or overlap syndrome) ii. drugs or toxins iii. Human Immunodeficiency Virus (HIV) infection iv. congenital heart defects repaired greater than 1 year prior to screening (i.e., atrial septal defects, ventricular septal defects, and patent ductus arteriosus) NB: subjects with portopulmonary hypertension and pulmonary veno-occlusive disease are NOT eligible for the study
* Subject must have a current diagnosis of being in World Health Organisation (WHO) Functional Class II or III.
* Subject must meet all of the following haemodynamic criteria by means of a right heart catheterization prior to screening:

  i. mPAP of ≥25 mmHg ii. PVR ≥ 300 dynes/sec/cm5 iii. PCWP or LVEDP of ≤12 mmHg if PVR ≥300 to <500 dyne/sec/cm5 , or PCWP/LVEDP ≤ 15 mmHg if PVR ≥500 dynes/sec/cm5
* Subject must walk a distance of ≥125m and ≤500m at the screening visit

Exclusion Criteria:

* Subject received previous PAH therapy (phosphodiesterase type 5 inhibitor (PDE5i), endothelin receptor antagonist (ERA), chronic prostanoid*) within 4 weeks prior to the screening visit (*Chronic prostanoid use is considered >7 days of treatment)
* Subject received ERA treatment (e.g., bosentan or sitaxentan) or PDE5i treatment (e.g. Sildenafil) at any time AND discontinued due to tolerance issues other than those associated with liver function abnormalities
* Subjects who have previously discontinued ambrisentan or tadalafil in either another clinical study or commercial product (Volibris/Letairis or Adcirca) for safety or tolerability reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2010-10-01; Primary Completion 2014-07-31 (Actual); Study Completion 2014-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (131):
- United States (53):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Kissimmee, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Weston, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Oakbrook Terrace, Illinois
  - GSK Investigational Site, Carmel, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Portland, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, New Hyde Park, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- Australia (6):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Chermside, Queensland
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Perth, Western Australia
- Austria (2):
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Vienna
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
- Canada (5):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Québec, Quebec
- France (11):
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Bron
  - GSK Investigational Site, La Tronche
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Saint-Pierre
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (16):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Löwenstein, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Giessen, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Greifswald, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Greece (3):
  - GSK Investigational Site, Alexandroupoli
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Thessaloniki
- Italy (5):
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Pisa, Tuscany
- Japan (4):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Netherlands (3):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Rotterdam
- Spain (12):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Toledo
  - GSK Investigational Site, Valencia
- Sweden (5):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Umeå
  - GSK Investigational Site, Uppsala
- United Kingdom (4):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Clydebank
  - GSK Investigational Site, London
  - GSK Investigational Site, Sheffield

REFERENCES:
- [Derived] Kuwana M, Blair C, Takahashi T, Langley J, Coghlan JG. Initial combination therapy of ambrisentan and tadalafil in connective tissue disease-associated pulmonary arterial hypertension (CTD-PAH) in the modified intention-to-treat population of the AMBITION study: post hoc analysis. Ann Rheum Dis. 2020 May;79(5):626-634. doi: 10.1136/annrheumdis-2019-216274. Epub 2020 Mar 11. PMID 32161055
- [Derived] White RJ, Vonk-Noordegraaf A, Rosenkranz S, Oudiz RJ, McLaughlin VV, Hoeper MM, Grunig E, Ghofrani HA, Chakinala MM, Barbera JA, Blair C, Langley J, Frost AE. Clinical outcomes stratified by baseline functional class after initial combination therapy for pulmonary arterial hypertension. Respir Res. 2019 Sep 12;20(1):208. doi: 10.1186/s12931-019-1180-1. PMID 31511080
- [Derived] Coghlan JG, Galie N, Barbera JA, Frost AE, Ghofrani HA, Hoeper MM, Kuwana M, McLaughlin VV, Peacock AJ, Simonneau G, Vachiery JL, Blair C, Gillies H, Miller KL, Harris JHN, Langley J, Rubin LJ; AMBITION investigators. Initial combination therapy with ambrisentan and tadalafil in connective tissue disease-associated pulmonary arterial hypertension (CTD-PAH): subgroup analysis from the AMBITION trial. Ann Rheum Dis. 2017 Jul;76(7):1219-1227. doi: 10.1136/annrheumdis-2016-210236. Epub 2016 Dec 30. PMID 28039187
- [Derived] Galie N, Barbera JA, Frost AE, Ghofrani HA, Hoeper MM, McLaughlin VV, Peacock AJ, Simonneau G, Vachiery JL, Grunig E, Oudiz RJ, Vonk-Noordegraaf A, White RJ, Blair C, Gillies H, Miller KL, Harris JH, Langley J, Rubin LJ; AMBITION Investigators. Initial Use of Ambrisentan plus Tadalafil in Pulmonary Arterial Hypertension. N Engl J Med. 2015 Aug 27;373(9):834-44. doi: 10.1056/NEJMoa1413687. PMID 26308684
- [Derived] Peacock AJ, Zamboni W, Vizza CD. Ambrisentan for the treatment of adults with pulmonary arterial hypertension: a review. Curr Med Res Opin. 2015;31(9):1793-807. doi: 10.1185/03007995.2015.1074890. Epub 2015 Aug 27. PMID 26196225

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 500 participants (par.) in the ITT Population were also included in the modified ITT Population (those who also met the modified inclusion/exclusion criteria defined in the protocol amendment 2). Disposition results below have been presented for the ITT Population.
Pre-assignment Details: A total of 610 par. were randomized; however, only 605 were included in the Intent-to-Treat (ITT) Population (randomized par. who received at least one dose of IP). All par. received a minimum of 24 weeks of therapy unless they died or withdrew.
Groups:
- Combination Therapy: Ambrisentan + Tadalafil: Participants initially received one tablet of 5 milligrams (mg) ambrisentan (AMB) and one tablet of AMB matching placebo once daily (QD) for the first 8 weeks plus one tablet of 20 mg tadalafil (TAD) and one tablet of TAD matching placebo QD for the first 4 weeks. The TAD dose was uptitrated to 40 mg (two tablets of 20 mg QD) after 4 weeks and the AMB dose may have been uptitrated to 10 mg (two tablets of 5 mg QD) after 8 weeks. The uptitration of AMB to 10 mg was not mandatory if the investigator decided for tolerability reasons the participants should remain on 5 mg.
- Ambrisentan Monotherapy: Participants initially received one tablet of 5 mg AMB and one tablet of AMB matching placebo QD for the first 8 weeks plus two tablets of TAD matching placebo. The AMB dose may have been uptitrated to 10 mg (two tablets of 5 mg QD) and two tablets of TAD matching placebo after 8 weeks. The uptitration of AMB to 10 mg was not mandatory if the investigator decided for tolerability reasons the participants should remain on 5 mg.
- Tadalafil Monotherapy: Participants initially received one tablet of 20 mg TAD and one tablet of TAD matching placebo QD for the first 4 weeks plus two tablets of AMB matching placebo. The TAD dose was uptitrated to 40 mg (two tablets of 20 mg QD) and two tablets of AMB matching placebo after 4 weeks.
Period: Overall Study
Arm/Group | Combination Therapy: Ambrisentan + Tadalafil | Ambrisentan Monotherapy | Tadalafil Monotherapy
Started | 302 | 152 | 151
Completed | 240 | 108 | 105
Not Completed | 62 | 44 | 46
Not completed — Adverse Event | 34 | 27 | 24
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 3
Not completed — Physician Decision | 14 | 10 | 10
Not completed — Withdrawal by Subject | 10 | 6 | 8
Not completed — Missing Completion Status | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy: Ambrisentan + Tadalafil | Ambrisentan Monotherapy | Tadalafil Monotherapy | Total
Number analyzed (Participants) | 302 | 152 | 151 | 605
Age, Continuous [Mean (Standard Deviation); unit: Years] — Intent-to-Treat Population
  Years | 55.9 (13.86) | 55.2 (14.41) | 55.9 (14.75) | 55.7 (14.21)
Sex: Female, Male [Count of Participants; unit: Participants] — Intent-to-Treat Population
  Participants
    Female | 223 | 117 | 121 | 461
    Male | 79 | 35 | 30 | 144
Race/Ethnicity, Customized [Number; unit: Participants] — Intent-to-Treat Population
  Participants
    African American/African Heritage | 11 | 14 | 13 | 38
    American Indian or Alaskan Native | 2 | 0 | 0 | 2
    Asian - Central/South Asian Heritage | 1 | 2 | 1 | 4
    Asian - Japanese Heritage | 3 | 0 | 1 | 4
    Asian - South East Asian Heritage | 1 | 2 | 1 | 4
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 3
    White - Arabic /North African Heritage | 1 | 1 | 0 | 2
    White - White/Caucasian/European Heritage | 280 | 131 | 133 | 544
    Mixed Race | 2 | 1 | 0 | 3
    Missing | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Adjudicated Clinical Failure (CF) Event, Death, Hospitalisation for Worsening PAH, Disease Progression, Unsatisfactory Long-term Clinical Response, All Through FAV
Description: Time to the first adjudicated CF event (death, hospitalization for worsening pulmonary arterial hypertension [PAH], disease progression, or unsatisfactory long-term clinical response) after initiating either first-line combination therapy with AMB and TAD or first-line monotherapy with either drug (AMB or TAD) in par. with PAH was assessed. If data was not available for some par. following a loss to follow-up, their event times were treated as censored at their last assessment time for the statistical analyses. FAV occurred approximately 4 weeks after the predicted 105th adjudicated first CF event was reached. Par. who had an FAV, and who had no adjudicated events or whose first adjudicated event occurred after their FAV, were censored at their individual FAV. Modified Intent-to-Treat (mITT) Population: all randomized par. who met the PAH diagnosis and inclusion/exclusion criteria defined in protocol amendment 2 and who also received at least one dose of investigational product (IP).
Time Frame: From Baseline up to the Final Assessment Visit (FAV) (average of 609 days)
Population: mITT Population
Measure: Number; unit: Participants
Groups:
- Monotherapy Pooled: Ambrisentan or Tadalafil: Participants initially received one tablet of 5 mg AMB and one tablet of AMB matching placebo QD for the first 8 weeks; or one tablet of 20 mg TAD and one tablet of TAD-matching placebo QD for the first 4 weeks. For participants on TAD, the dose of TAD was uptitrated to 40 mg (two tablets of 20 mg QD) after 4 weeks and for participants on AMB, the dose of AMB may have been uptitrated to 10 mg (two tablets of 5 mg QD) after 8 weeks. The uptitration of AMB to 10 mg was not mandatory if the investigator decided for tolerability reasons the participants should remain on 5 mg.
Arm/Group | Combination Therapy: Ambrisentan + Tadalafil | Monotherapy Pooled: Ambrisentan or Tadalafil | Ambrisentan Monotherapy | Tadalafil Monotherapy
Number analyzed (Participants) | 253 | 247 | 126 | 121
Participants
  First adjudicated clinical failure event | 46 | 77 | 43 | 34
  Death (all-cause) | 9 | 8 | 2 | 6
  Hospitalization for worsening PAH | 10 | 30 | 18 | 12
  Disease progression | 10 | 16 | 12 | 4
  Unsatisfactory long-term clinical response | 17 | 23 | 11 | 12
Statistical Analysis 1: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Monotherapy Pooled: Ambrisentan or Tadalafil; Test type: Superiority or Other; p = 0.0002, Stratified Log Rank; Hazard Ratio (HR) = 0.502, 95% CI 2-sided [0.348 to 0.724] — Analysis of time to first adjudicated clinical failure event through FAV. HR is calculated using the Cox proportional hazards model. HR is for Combination Therapy: Ambrisentan + Tadalafil / Monotherapy Pooled: Ambrisentan or Tadalafil
Statistical Analysis 2: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Ambrisentan Monotherapy; Test type: Superiority or Other; p = 0.0004, Stratified Log Rank; Hazard Ratio (HR) = 0.477, 95% CI 2-sided [0.314 to 0.723] — Analysis of time to first adjudicated clinical failure event through FAV. HR is calculated using the Cox proportional hazards model. HR is for Combination Therapy: Ambrisentan + Tadalafil / Ambrisentan Monotherapy
Statistical Analysis 3: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Tadalafil Monotherapy; Test type: Superiority or Other; p = 0.0045, Stratified Log Rank; Hazard Ratio (HR) = 0.528, 95% CI 2-sided [0.338 to 0.827] — Analysis of time to first adjudicated clinical failure event through FAV. HR is calculated using the Cox proportional hazards model. HR is for Combination Therapy: Ambrisentan + Tadalafil / Tadalafil Monotherapy

2. Secondary Outcome: Percent Change From Baseline in the N-Terminal Pro-B-Type Natriuretic Peptide at Week 24
Description: N-Terminal Pro-B-Type Natriuretic Peptide (NT-proBNP) is a surrogate marker of heart failure. The data were log-transformed. The geometric mean was calculated (based on the log-transformed data). The geometric mean ratio was calculated as the ratio between the Week 24 value and the Baseline value (based on the log-transformed data) and presented as percent change = 100 * (geometric mean ratio - 1). The Baseline value is the last value prior to administration of study drug; this may be prior to or on the day of study drug initiation. No imputation was performed for missing data. The secondary endpoints were analyzed according to a pre-specified hierarchical testing procedure.
Time Frame: Baseline and Week 24
Population: mITT Population. Only participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Combination Therapy: Ambrisentan + Tadalafil | Monotherapy Pooled: Ambrisentan or Tadalafil | Ambrisentan Monotherapy | Tadalafil Monotherapy
Number analyzed (Participants) | 204 | 199 | 99 | 100
Percent change | -67.15 (0.069) | -50.37 (0.070) | -56.15 (0.096) | -43.83 (0.095)
Statistical Analysis 1: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Monotherapy Pooled: Ambrisentan or Tadalafil; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Percent Difference = -33.81, 95% CI 2-sided [-44.78 to -20.66] — Mean percent difference is for Combination Therapy: Ambrisentan + Tadalafil - Monotherapy Pooled: Ambrisentan or Tadalafil
Statistical Analysis 2: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Ambrisentan Monotherapy; Test type: Superiority or Other; p = 0.0111, ANCOVA; Mean Percent Difference = -25.09, 95% CI 2-sided [-40.04 to -6.40] — Mean percent difference is for Combination Therapy: Ambrisentan + Tadalafil - Ambrisentan Monotherapy
Statistical Analysis 3: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Tadalafil Monotherapy; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Percent Difference = -41.51, 95% CI 2-sided [-53.16 to -26.97] — Mean percent difference is for Combination Therapy: Ambrisentan + Tadalafil - Tadalafil Monotherapy

3. Secondary Outcome: Percentage of Participants With a Satisfactory Clinical Response at Week 24
Description: A satisfactory clinical response at Week 24 is defined as a participant who meets all of the following criteria: 10% improvement in 6MWD compared with Baseline; improvement to or maintenance of World Health Organization (WHO) class I or II symptoms; no events of clinical worsening prior to or at the Week 24 visit. Clinical worsening events included: death, hospitalization for pulmonary arterial hypertension (PAH), and disease progression. Participants without an event of clinical worsening prior to or at the Week 24 visit who did not have a 6MWD value or a WHO functional class value at Week 24 were excluded from the analysis.
Time Frame: Baseline and Week 24
Population: mITT Population. Only those participants who had a "Yes"/"No" response were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Combination Therapy: Ambrisentan + Tadalafil | Monotherapy Pooled: Ambrisentan or Tadalafil | Ambrisentan Monotherapy | Tadalafil Monotherapy
Number analyzed (Participants) | 234 | 226 | 113 | 113
Percentage of participants | 39 | 29 | 31 | 27
Statistical Analysis 1: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Monotherapy Pooled: Ambrisentan or Tadalafil; Test type: Superiority or Other; p = 0.0264, Regression, Logistic; Odds Ratio (OR) = 1.563, 95% CI 2-sided [1.054 to 2.319] — Odds ratio is for Combination Therapy: Ambrisentan + Tadalafil / Monotherapy Pooled: Ambrisentan or Tadalafil
Statistical Analysis 2: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Ambrisentan Monotherapy; Test type: Superiority or Other; p = 0.1518, Regression, Logistic; Odds Ratio (OR) = 1.424, 95% CI 2-sided [0.878 to 2.308] — Odds ratio is for Combination Therapy: Ambrisentan + Tadalafil / Ambrisentan Monotherapy
Statistical Analysis 3: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Tadalafil Monotherapy; Test type: Superiority or Other; p = 0.0321, Regression, Logistic; Odds Ratio (OR) = 1.723, 95% CI 2-sided [1.047 to 2.833] — Odds ratio is for Combination Therapy: Ambrisentan + Tadalafil / Tadalafil Monotherapy

4. Secondary Outcome: Change From Baseline in the 6 Minute Walk Distance Test at Week 24
Description: The 6-minute walk distance (6MWD) test measures the distance that a participant can walk in a period of 6 minutes. Change from Baseline was calculated as the Week 24 value minus the Baseline value. The analysis was performed based on last observation carried forward data, except in the case of an adjudicated clinical failure event of death or hospitalization preceding the missing data observation. In this case, the missing observation was assigned the worst-rank score relative to those actually observed and was assigned a rank reflecting the relative order of the actual event times. Baseline 6MWD comprised of an average of the last two consecutive measurements prior to randomization that varied by no greater than 10%. If only one measurement was available, that measurement was used. If no two consecutive measures vary by no greater than 10% then Baseline was based on the last two consecutive measures for a participant.
Time Frame: Baseline and Week 24
Population: mITT Population. Only participants with Baseline data were analyzed.
Measure: Median (95% Confidence Interval); unit: Meters
Arm/Group | Combination Therapy: Ambrisentan + Tadalafil | Monotherapy Pooled: Ambrisentan or Tadalafil | Ambrisentan Monotherapy | Tadalafil Monotherapy
Number analyzed (Participants) | 248 | 244 | 124 | 120
Meters | 48.98 [39.00 to 57.50] | 23.80 [19.00 to 33.50] | 27.00 [12.50 to 38.00] | 22.70 [16.50 to 35.50]
Statistical Analysis 1: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Monotherapy Pooled: Ambrisentan or Tadalafil; Test type: Superiority or Other; p < 0.0001, Stratified Wilcoxon Rank Sum Test; Median Difference = 22.75, 95% CI 2-sided [12.00 to 33.50] — Median difference is for Combination Therapy: Ambrisentan + Tadalafil - Monotherapy Pooled: Ambrisentan or Tadalafil
Statistical Analysis 2: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Ambrisentan Monotherapy; Test type: Superiority or Other; p = 0.0005, Stratified Wilcoxon Rank Sum Test; Median Difference = 24.75, 95% CI 2-sided [11.00 to 38.50] — Median difference is for Combination Therapy: Ambrisentan + Tadalafil - Ambrisentan Monotherapy
Statistical Analysis 3: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Tadalafil Monotherapy; Test type: Superiority or Other; p = 0.0030, Stratified Wilcoxon Rank Sum Test; Median Difference = 20.85, 95% CI 2-sided [8.00 to 33.70] — Median difference is for Combination Therapy: Ambrisentan + Tadalafil - Tadalafil Monotherapy

5. Secondary Outcome: Change From Baseline in the World Health Organization Functional Class at Week 24
Description: The WHO Functional Class (FC) indicates the severity of PAH and is an adaptation of the New York Heart Association classification. It was assessed by the investigator. There are four grades for WHO FC based on severity of symptoms (Class I = none, Class IV = most severe). Baseline WHO FC is the latest assessment prior to dosing (i.e., at Randomization or Screening). Change from Baseline at Week 24 was calculated as the Week 24 value minus the Baseline value. The analysis was performed based on the last observation carried forward data, except in the case of an adjudicated clinical failure event of death or hospitalization preceding the missing data observation. In this case, the missing observations was assigned the worst-rank score relative to those actually observed and was assigned rank reflecting the relative order of the actual event times.
Time Frame: Baseline and Week 24
Population: mITT Population. Only participants with Baseline data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Combination Therapy: Ambrisentan + Tadalafil | Monotherapy Pooled: Ambrisentan or Tadalafil | Ambrisentan Monotherapy | Tadalafil Monotherapy
Number analyzed (Participants) | 252 | 244 | 124 | 120
Scores on a scale | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0] | 0.0 [-1.0 to 0.0]
Statistical Analysis 1: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Monotherapy Pooled: Ambrisentan or Tadalafil; Test type: Superiority or Other; p = 0.2287, Stratified Wilcoxon Rank Sum Test; Median Difference = 0.0, 95% CI 2-sided [0.0 to 0.0] — Median difference is for Combination Therapy: Ambrisentan + Tadalafil - Monotherapy Pooled: Ambrisentan or Tadalafil
Statistical Analysis 2: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Ambrisentan Monotherapy; Test type: Superiority or Other; Stratified Wilcoxon Rank Sum Test; This comparison was not formally tested according to the pre-defined hierarchical testing procedure; Median Difference = 0.0, 95% CI 2-sided [0.0 to 0.0] — Median difference is for Combination Therapy: Ambrisentan + Tadalafil - Ambrisentan Monotherapy
Statistical Analysis 3: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Tadalafil Monotherapy; Test type: Superiority or Other; Stratified Wilcoxon Rank Sum Test; This comparison was not formally tested according to the pre-defined hierarchical testing procedure; Median Difference = 0.0, 95% CI 2-sided [0.0 to 0.0] — Median difference is for Combination Therapy: Ambrisentan + Tadalafil - Tadalafil Monotherapy

6. Secondary Outcome: Change From Baseline in Borg Dyspnea Index at Week 24
Description: Borg Dyspnea Index (BDI) indicates the degree of breathlessness after completion of the 6 minute walk test. The BDI was calculated by using the Borg category (C) ratio (R) CR10 scale which starts at 0 (nothing at all) and has no upper limit (extremely strong). Change from BL was calculated as the Week 24 values minus the BL value. The BDI scale was assessed by each participant. The BL BDI score is the average of the two BDI values obtained following the two 6MWD tests used in determining the BL 6MWD. A negative change from BL in the BDI score represented an improvement for the participant. The analysis was performed based on the last observation carried forward data, except in the case of an adjudicated clinical failure event of death or hospitalization preceding the missing data observation. In this case, the missing observation was assigned the worst-rank score relative to those actually observed and was assigned rank reflecting the relative order of the actual event times.
Time Frame: Baseline (BL) and Week 24
Population: mITT Population. Only participants with Baseline data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Combination Therapy: Ambrisentan + Tadalafil | Monotherapy Pooled: Ambrisentan or Tadalafil | Ambrisentan Monotherapy | Tadalafil Monotherapy
Number analyzed (Participants) | 247 | 244 | 124 | 120
Scores on a scale | -1.00 [-2.00 to 0.50] | -0.50 [-1.50 to 0.50] | -0.50 [-1.50 to 0.50] | -0.50 [-2.00 to 0.88]
Statistical Analysis 1: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Monotherapy Pooled: Ambrisentan or Tadalafil; Test type: Superiority or Other; Stratified Wilcoxon Rank Sum Test; This endpoint was not formally tested according to the pre-defined hierarchical testing procedure; Median Difference = -0.38, 95% CI 2-sided [-0.75 to 0.00] — Median difference is for Combination Therapy: Ambrisentan + Tadalafil - Monotherapy Pooled: Ambrisentan or Tadalafil
Statistical Analysis 2: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Ambrisentan Monotherapy; Test type: Superiority or Other; Stratified Wilcoxon Rank Sum Test; This endpoint was not formally tested according to the pre-defined hierarchical testing procedure; Median Difference = -0.50, 95% CI 2-sided [-1.00 to 0.00] — Median difference is for Combination Therapy: Ambrisentan + Tadalafil - Ambrisentan Monotherapy
Statistical Analysis 3: Comparison: Combination Therapy: Ambrisentan + Tadalafil vs Tadalafil Monotherapy; Test type: Superiority or Other; Stratified Wilcoxon Rank Sum Test; This endpoint was not formally tested according to the pre-defined hierarchical testing procedure; Median Difference = -0.50, 95% CI 2-sided [-1.00 to 0.00] — Median difference is for Combination Therapy: Ambrisentan + Tadalafil - Tadalafil Monotherapy

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of investigational product until 30 days after the last dose of investigational product (average of 639 days on investigational product).
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all randomized participants who received at least one dose of investigational product. Only AEs for the "On-Randomized Treatment" arms are tabulated.
Arm/Group | Combination Therapy: Ambrisentan + Tadalafil | Ambrisentan Monotherapy | Tadalafil Monotherapy
Serious Adverse Events (participants affected / at risk) | 124/302 | 63/152 | 68/151
Other Adverse Events (participants affected / at risk) | 279/302 | 140/152 | 135/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy: Ambrisentan + Tadalafil (N=302) | Ambrisentan Monotherapy (N=152) | Tadalafil Monotherapy (N=151)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 11 | 16 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary vasculitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 15 | 10 | 7
Respiratory tract infection (Infections and infestations) | 4 | 1 | 1
Lung infection (Infections and infestations) | 3 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 5 | 3
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 1
Abscess limb (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 3
Catheter site infection (Infections and infestations) | 1 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways diseas (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 3
Septic shock (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Alveolar osteitis (Infections and infestations) | 0 | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 1 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
West Nile viral infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 6 | 6 | 3
Right ventricular failure (Cardiac disorders) | 5 | 8 | 3
Atrial flutter (Cardiac disorders) | 3 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 2 | 1
Angina pectoris (Cardiac disorders) | 2 | 2 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 2
Coronary artery stenosis (Cardiac disorders) | 2 | 0 | 0
Supraventricular tachyarrhythmia (Cardiac disorders) | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 3
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0 | 0
Cor pulmonale acute (Cardiac disorders) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pleuropericarditis (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1
Cardiorenal syndrome (Cardiac disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 7 | 0 | 0
Oedema peripheral (General disorders) | 5 | 1 | 0
Pyrexia (General disorders) | 4 | 1 | 1
Death (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 2
Drug withdrawal syndrome (General disorders) | 0 | 1 | 0
Euthanasia (General disorders) | 0 | 0 | 1
Infusion site phlebitis (General disorders) | 0 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 3 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 1 | 0 | 0
Epiploic appendagitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 10 | 3 | 5
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0 | 0
Hyperchromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 9 | 5 | 7
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 2 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 5 | 1 | 4
Fluid retention (Metabolism and nutrition disorders) | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon adenoma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Mountain sickness acute (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 1
Transaminases increased (Investigations) | 2 | 0 | 0
Blood pressure systolic increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 3 | 2 | 2
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 1 | 0
Vascular insufficiency (Vascular disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1
Diabetes insipidus (Endocrine disorders) | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Autoimmune disorder (Immune system disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy: Ambrisentan + Tadalafil (N=302) | Ambrisentan Monotherapy (N=152) | Tadalafil Monotherapy (N=151)
Oedema peripheral (General disorders) | 133 | 60 | 44
Fatigue (General disorders) | 35 | 22 | 20
Non-cardiac chest pain (General disorders) | 26 | 14 | 9
Pyrexia (General disorders) | 17 | 6 | 2
Chest discomfort (General disorders) | 16 | 6 | 5
Asthenia (General disorders) | 9 | 4 | 8
Pain (General disorders) | 8 | 2 | 8
Nasopharyngitis (Infections and infestations) | 51 | 32 | 24
Upper respiratory tract infection (Infections and infestations) | 41 | 23 | 22
Bronchitis (Infections and infestations) | 34 | 7 | 10
Urinary tract infection (Infections and infestations) | 24 | 12 | 18
Sinusitis (Infections and infestations) | 22 | 11 | 11
Influenza (Infections and infestations) | 14 | 9 | 7
Headache (Nervous system disorders) | 124 | 51 | 55
Dizziness (Nervous system disorders) | 62 | 31 | 22
Presyncope (Nervous system disorders) | 11 | 6 | 11
Syncope (Nervous system disorders) | 9 | 4 | 8
Diarrhoea (Gastrointestinal disorders) | 63 | 35 | 26
Nausea (Gastrointestinal disorders) | 47 | 23 | 23
Vomiting (Gastrointestinal disorders) | 35 | 13 | 13
Dyspepsia (Gastrointestinal disorders) | 32 | 6 | 18
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 23 | 10 | 15
Constipation (Gastrointestinal disorders) | 17 | 10 | 6
Abdominal pain (Gastrointestinal disorders) | 9 | 9 | 7
Abdominal pain upper (Gastrointestinal disorders) | 8 | 6 | 8
Dry mouth (Gastrointestinal disorders) | 8 | 11 | 3
Abdominal distension (Gastrointestinal disorders) | 4 | 8 | 11
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 58 | 25 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 53 | 20 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 | 27 | 28
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27 | 7 | 15
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 18 | 9 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 9 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 49 | 16 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 43 | 17 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 | 21 | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 30 | 12 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 25 | 8 | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 10 | 4 | 8
Flushing (Vascular disorders) | 41 | 18 | 15
Hypotension (Vascular disorders) | 21 | 8 | 9
Anaemia (Blood and lymphatic system disorders) | 38 | 8 | 11
Insomnia (Psychiatric disorders) | 21 | 6 | 10
Depression (Psychiatric disorders) | 13 | 3 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 8 | 5
Fluid retention (Metabolism and nutrition disorders) | 16 | 7 | 9
Decreased appetite (Metabolism and nutrition disorders) | 10 | 9 | 8
Rash (Skin and subcutaneous tissue disorders) | 24 | 6 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 10 | 6
Palpitations (Cardiac disorders) | 33 | 22 | 20
Vision blurred (Eye disorders) | 19 | 8 | 4
Vertigo (Ear and labyrinth disorders) | 5 | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.